CLINICAL TRIAL: NCT04705870
Title: Comparison of the Performance of an Optimized 3D EPI SWI Sequence and a Non-EPI QSM SWI Sequence in Detecting the Central Vein Sign in Patients With Multiple Sclerosis
Acronym: COPEQ-MS
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2020_39
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cerebral MRI — MRI of routine care in the context of MS includes at least the following sequences:
  * 3D T1 TFE (2 minutes)
  * T2 TSE (2 minutes)
  * 3D FLAIR (3 minutes)
  * SWI EPI 0.6 iso (7 minutes)
  The sequences added by the search are:
  * SWI non EPI QSM 6 echo (10 minutes)
  * SWI EPI in resolution equivalent to non-EPI SWI (3 minutes)
  * SWI EPI to TR equivalent to SWI non EPI (6 minutes)

SUMMARY:
Patients who have agreed to participate in the study will complete the MRI protocol as part of routine care, to which four additional 20-minute sequences will be added.

MRI of routine care in the context of MS includes at least the following sequences:

* 3D T1 TFE (2 minutes)
* T2 TSE (2 minutes)
* 3D FLAIR (3 minutes)
* SWI EPI 0.6 iso (7 minutes)

The sequences added by the search are:

* SWI non EPI QSM 6 echo (10 minutes)
* SWI EPI in resolution equivalent to non-EPI SWI (3 minutes)
* SWI EPI to TR equivalent to SWI non EPI (6 minutes)

These sequences will be acquired before or after the injection of gadolinium (if present in the examination of routine care). For examinations carried out with injection, the order of carrying out the 4 post-injection SWI sequences will be random.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* With MS defined according to the McDonald's revised clinical or radiological spatial and temporal dissemination criteria, with onset of symptoms <5 years
* To benefit as part of care from an MRI with or without injection of gadolinium
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with MS and who should undergo an MRI examination with or without injections of contrast agent as part of their care.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
percentage of lesions showing the central vein sign with the SWI EPI sequence that also show the central vein sign with the candidate sequence | 1 day
percentage of lesions which do not present the sign of the central vein with the SWI EPI sequence but which present it with the candidate sequence | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Hhopital fondation adolphe de rothschild, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No